CLINICAL TRIAL: NCT04701229
Title: Impact of the Double Haploinsufficiency of the RBM22 and SLU7 Genes in Del(5q) Myelodysplastic Syndromes Isolated or Not Compared to the Single Haploinsufficiency of RBM22 and Normal Karyotype Myelodysplastic Syndromes.
Brief Title: Haploinsufficiency of the RBM22 and SLU7 Genes in Del(5q) Myelodysplastic Syndromes
Acronym: SMD-RMB22
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: SMD-RMB22 (29BRC20.0029)
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Myelodysplastic Syndromes; Myelodysplastic Syndrome With Isolated Del(5Q); Myelodysplastic Syndrome With Del(5Q)
Keywords: RBM22; SLU7; transformation to acute myeloid leukemia; anemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Chromosome 5q Deletion Syndrome; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — cytogenetic pellets; bone marrow patients cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- normal karyotype: control group
  Interventions: Genetic: somatic cytogenetic and genetic characterization
- del5q-RBM22neg-SLU7neg: this group is characterized by its karyotype. It presents a 5q deletion, a loss of RBM22, a loss of SLU7.
  Interventions: Genetic: somatic cytogenetic and genetic characterization
- del5q-RBM22neg-SLU7pos: this group is characterized by its karyotype. It presents a 5q deletion, a loss of RBM22 but no loss of SLU7
  Interventions: Genetic: somatic cytogenetic and genetic characterization
- del5q-RBM22pos-SLU7neg: this group is characterized by its karyotype. It presents a 5q deletion, and no loss of RBM22, but a loss in SLU7
  Interventions: Genetic: somatic cytogenetic and genetic characterization
- del5q-RBM22pos-SLU7pos: this group is characterized by its karyotype. It presents a 5q deletion, and no loss of RBM22 nor SLU7
  Interventions: Genetic: somatic cytogenetic and genetic characterization

INTERVENTIONS:
Genetic: somatic cytogenetic and genetic characterization — investigating the presence of some genes allelles (RBM22, SLU7, RBM27, other on chromosome 5) by FISH, and sequencing of a classical panel of myeloid genes including RBM22, SLU7, for somatic identification of genetic alterationss of the blasts.

SUMMARY:
Myelodysplastic syndromes (MDS) are malignant hematopathies of the elderly characterized by persistent cytopenias and the presence of deregulated clonal hematopoiesis. The risk of progression to acute myeloid leukemia (AML) is variable. Acquired cytogenetic abnormalities are found in less than 50% of de novo cases and up to 80% in secondary MDS. The deletion of the long arm of chromosome 5 (written del(5q)) is the most common abnormality in MDS (15%). Del(5q) MDS has a good prognosis, with a median survival of 6 years and a 15% risk of progression to AML. However, their life expectancy is shorter than the general population, and the quality of life of patients is diminished. These treatments are not that effective over a long period of time or not well tolerated, and the majority of patients die from causes related to their MDS, such as infections (38%), progression to AML (15%), or bleeding (13%). Two genes, RBM22 and SLU7, coding for proteins of the same complex involved in splicing pre-messenger RNA are carried on the long arm of chromosome 5. We investigate the pronostic impact and the predictive value of the double haploinsufficiency of the RBM22 and SLU7 genes in del(5q) myelodysplastic syndromes isolated or not compared to the single haploinsufficiency of RBM22 and normal karyotype myelodysplastic syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with del5q MDS isolated or not
* The clinical and biological data are known at the time of diagnosis.
* The clinical and biological data are known 1 year after the diagnosis
* Consent for the collection of samples for research purposes
* Non-opposition obtained

Exclusion Criteria:

* Patients under judicial protection (guardianship, ...)
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with myelodysplastic syndromes and presenting a deletion of chromosome 5 in their bone marrow cells
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
prognostic impact on anemia | retrospective study on data collected; 2 years
  To evaluate the prognostic impact of the dual loss of an RBM22 and a SLU7 allele compared to the loss of an RBM22 allele alone on anemia, as measured by the hemoglobin level in the blood, between diagnosis and one year in patients with del5q myelodysplastic syndrome.

SECONDARY OUTCOMES:
prognostic impact on blood count | retrospective study on data collected; 2 years
  To evaluate the prognostic impact of the double loss of an RBM22 allele and a SLU7 allele compared to the loss of an RBM22 allele alone on the other criteria of the blood count including leukocytes, platelets, monocytes, circulating blasts, VGM, myelemia.
prognostic impact on progression to leukemia | retrospective study on data collected; 2 years
  To evaluate the prognostic impact of the double loss of an RBM22 and a SLU7 allele compared to the loss of an RBM22 allele alone on the progression to acute myeloid leukemia.
impact on gene expression and splicing profile | retrospective study on RNA collected; 2 years
  To evaluate the impact of the double loss of an RBM22 allele and a SLU7 allele compared to the loss of an RBM22 allele alone on gene expression profiles, including splicing variants.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Bérengère TROADEC, Principal Investigator — CHRU Brest
Locations (3):
- France (3):
  - CHRU de Brest, Brest
  - Groupe Français de cytogénétique Hématologique, Paris
  - Groupe Français des Myélodysplasies, Paris

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.